CLINICAL TRIAL: NCT02613065
Title: The Role of Protein in Regulating Ad Libitum Energy Intake in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Principal Investigator, David Allison, Phd, School of Public Health Associate Dean for Research, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: F141121006
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Energy Balance
Keywords: Ad libitum; Energy balance; Protein

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eggwhite protein shake (Experimental): Participants drink a NOW Foods protein shake (~20% daily energy requirements) at the beginning of each of the three daily meals. Kcals/meal are dependent upon participant's baseline Resting Metabolic Rate value.
  Interventions: Dietary Supplement: Consumption of NOW Foods eggwhite protein shake
- Maltodextrin carbohydrate shake (Active Comparator): Participants drink a NOW Foods carbohydrate shake (~20% daily energy requirements) at the beginning of each of the three daily meals. Kcals/meal are dependent upon participant's baseline Resting Metabolic Rate value.
  Interventions: Dietary Supplement: Consumption of NOW Foods maltodextrin shake

INTERVENTIONS:
Dietary Supplement: Consumption of NOW Foods eggwhite protein shake — Consumption of NOW Foods egg white protein shake at beginning of 3 daily meals that in total, is approximately 20% of caloric needs.
  Arms: Eggwhite protein shake
Dietary Supplement: Consumption of NOW Foods maltodextrin shake — Consumption of NOW Foods maltodextrin shake at beginning of 3 daily meals that in total, is approximately 20% of caloric needs.
  Arms: Maltodextrin carbohydrate shake

SUMMARY:
The purpose of this project is to determine if protein is less likely to create positive energy balance when added to the diet compared to carbohydrate. To do this, the investigators will take detailed measurements of participant's baseline metabolic rate to understand their energy requirements. Then, the investigators will feed participants all their meals for two weeks, Monday-Friday, and measure their food intake. During one of the week-long feeding periods, participants will consume a shake made of egg protein that is ~20% of their energy requirements. During the other week, participants will consume a shake made of carbohydrate that is ~20% of their energy requirements. Participants will drink the assigned shake at the beginning of each of their daily three meals, and then they will be offered a 'regular' meal of unlimited quantity. Participants will not know that the investigators are measuring the food consumed after drinking the shake. Participants will drink the protein shake for the first week and carb-based shake for the second week, and vice versa-- depending on the randomization order. To account for energy expenditure, participants will wear an activity monitor, an accelerometer. Energy balance, measured as participant energy intake minus energy expenditure, will be our main outcome for each treatment. However, because participants may change their behavior if made aware of the true research question, the investigators will tell participants that the purpose of the study is to see how low fiber and high fiber shakes affect mood. The hypothesis is that during the week when participants consume the protein shake, they will remain in energy balance, but during the week of carbohydrate shake consumption, participants will have positive energy balance.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥20, and ≤30 kg/m2
* Moderately active or sedentary (Physical Activity Level <2.0)

Exclusion Criteria:

* Any food allergy.
* Religious affiliations that include specific food guidelines.
* Participation in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months.
* Weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss.
* Currently taking medication that suppresses or stimulates appetite or that affects body weight, including oral anti-diabetic medications.
* History of prior surgical procedure for weight control.
* Anyone currently taking statins.
* Claustrophobia
* Current smoker or quit smoking less than 6 months prior.
* Any major disease, including:
* Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
* Active or chronic infections, including self-reported HIV positivity and active tuberculosis. -Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months.
* Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Active renal disease.
* Lung disease: chronic obstructive airway disease requiring use of oxygen.
* Diagnosed diabetes (type 1 or 2).
* Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.
* A score on the Brief Symptom Inventory (BSI) (Derogatis & Melisaratos, 1983) that exceeds the 90th percentile.
* History of or current eating disorders, or an Eating Attitudes Test (EAT-26) score >20.
* Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; another household member is a participant or staff member in the trial; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating clinics before trial completed; unable to walk 0.25 mile in 10 minutes.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months.
* A recent or ongoing problem with drug abuse or addiction.
* Excessive alcohol intake, either acute or chronic, defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months; or 3) other evidence available to clinic staff.
* Pregnancy and childbearing: currently pregnant or less than 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the course of the trial; unwilling to take adequate contraceptive measures if potentially fertile.
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Energy Balance measured as participant energy intake (food weight before and after meals) minus energy expenditure (accelerometer) | 10 days
  Feeding periods are separated by two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David B Allison, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Gibson MJ, Dawson JA, Wijayatunga NN, Ironuma B, Chatindiara I, Ovalle F, Allison DB, Dhurandhar EJ. A randomized cross-over trial to determine the effect of a protein vs. carbohydrate preload on energy balance in ad libitum settings. Nutr J. 2019 Nov 9;18(1):69. doi: 10.1186/s12937-019-0497-4. PMID 31706311